CLINICAL TRIAL: NCT03807128
Title: MYeloma Resistance And Clonal Evolution
Acronym: MYRACLE
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0197; IDRCB - ANSM (Other: 2018-A01578-47)
Record Dates: First submitted 2018-09-26; First posted 2019-01-16 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Cohort; Resistance; Quality of life
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MYRACLE patients
  Interventions: Other: Prélèvement sanguin (2*4mL) ou médullaire (2mL); Other: Data collection through questionnaires

INTERVENTIONS:
Other: Prélèvement sanguin (2*4mL) ou médullaire (2mL) — Additional blood (2*4mL) or bone marrow (2mL) sample depending on clinical presentation of disease
Other: Data collection through questionnaires — Collection of quality of life and occupational exposure data via questionnaires

SUMMARY:
Multiple Myeloma (MM) is often associated with progression, temporary response to therapy and a high relapse rate over time resulting in a poor long-term prognosis. Because MM is classified as an incurable disease, therapeutic resistance is of great interest. However, knowledge about the biological mechanisms underlying resistance associated with MM therapies and about associated predictors remains poor. The MYRACLE cohort, a multicenter prospective cohort of patients with MM, is set up to address this limitation.

DETAILED DESCRIPTION:
The MYRACLE cohort study aims at including all patients (>18 years old) who are diagnosed with MM in any stage of the disease and treated in specialized oncology centers in 2 public hospitals in Northwestern France. Any such patient providing a signed informed consent is included. All subjects are followed up until refusal to participate in the study, emigration or death. The MYRACLE follow-up is continuous and collects data on socio-economic status, medical status, MM therapies and associated events (resistance, side effects). Participants also complete standardized quality of life (QOL) questionnaires. In addition, participants are asked to donate blood samples that will support ex vivo analysis of expression and functional assays required to uncover predictive biomarkers and companion diagnostics. If diagnostic biopsies are performed during the course of the disease, extracted biological samples are kept in a dedicated biobank.

ELIGIBILITY:
Inclusion Criteria:

* Patient consulting due to the discovery or recurrence of MM according to international diagnostic criteria (IMWG 2014)
* Patient having consented to participate in the study and his/her biocollection
* Patient affiliated to or benefiting from a social security scheme or similar

Exclusion Criteria:

* Minors
* Major under guardianship or curatorship
* Protected persons.
* Pregnant or breast-feeding women
* Persons benefiting from the AME

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to multiple myeloma patients managed in the hematology departments of the University Hospital of Nantes and the CHD of La Roche sur Yon.
  Recruitment of the hematology departments of the University Hospital of Nantes and CHD of La Roche sur Yon makes it possible to envisage an annual recruitment of 60 new myeloma diagnoses, and an annual number of 80 relapses. These data are estimated from the number of files submitted to the Multidisciplinary Collaborative Meeting (RPN) and the annual inclusion number in clinical trials. This number represents a cohort of about 140 inclusions per year. The average number of visits can be estimated at 1.5 / year per patient.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2034-02-11 (Estimated); Study Completion 2049-02-11 (Estimated)

PRIMARY OUTCOMES:
Describe the mechanisms of resistance of myeloma cells. | 15 years
  Number of resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille TOUZEAU, PU, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - La Roche sur Yon Hospital Departmental, La Roche-sur-Yon
  - Nantes University Hospital, Nantes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Derrien J, Gastineau S, Frigout A, Giordano N, Cherkaoui M, Gaborit V, Boinon R, Douillard E, Devic M, Magrangeas F, Moreau P, Minvielle S, Touzeau C, Letouze E. Acquired resistance to a GPRC5D-directed T-cell engager in multiple myeloma is mediated by genetic or epigenetic target inactivation. Nat Cancer. 2023 Nov;4(11):1536-1543. doi: 10.1038/s43018-023-00625-9. Epub 2023 Aug 31. PMID 37653140